CLINICAL TRIAL: NCT03379116
Title: A Study on Nutrition Support in Adult Patients With Severe Burns
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, chief, Southeast University, China
Other Study IDs: 20171215
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Severe Burn; Enternal Nutrition
MeSH Terms: conditions — Burns | interventions — Enteral Nutrition; Parenteral Nutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: enteral nutrition and parenteral nutrition — In the treatment of the burned patients injured,data on nutritional support and patient's outcomes were collected and analyzed.

SUMMARY:
To delineate nutritional support in adults patients with severe burns to investigate associations between nutritional practice and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients were at least 18 years of age
* Patients were expected to survive more than 48 hours.

Exclusion Criteria:

* irreversible disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was a prospective, observational, multicenter trial and was conducted in intensive care units of seven hospitals participating in the treatment of the burn patients. Patients who were at least 18 years of age were eligible if they were expected to survive more than 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-06-02 (Actual); Primary Completion 2014-09-24 (Actual); Study Completion 2014-10-02 (Actual)

PRIMARY OUTCOMES:
Mortality at 28 days | 28days
  Daily data were recorded for a maximum of 28 days per patient. Patients alive in hospital at the 28th day or discharged prior to 28 days were considered to be survivors.